CLINICAL TRIAL: NCT04153279
Title: A Pilot Study of CMV-TCR-T Cells in CM Virus Infection Diseases After HSCT
Brief Title: CMV-TCR-T Cells for CM Virus Infection After HSCT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hebei Yanda Ludaopei Hospital (Other)
Collaborators: China Immunotech (Beijing) Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HXYT-005
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-11

CONDITIONS: CMV Infection or Reactivation After Allogenic HSCT
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CMV-TCR-T cells (Experimental): The patients will receive one dose of CMV-TCR-T.The dosage ranges from 0.1×10^6 to 1×10^6 TCR+T/Kg.
  Interventions: Biological: CMV-TCR-T cells

INTERVENTIONS:
Biological: CMV-TCR-T cells — Patients with CMV emias or CMV disease will be enrolled, and donor derived CMV-TCR-T(HLA-A*1101\0201\2402) cells will be intravenously infused with a escalated dose of 0.1-1×106 CMV-TCR-T cells. The CMV DNA copies and CMV-TCR-T cell proliferation will be monitored in the scheduled time (day 0, day 4, day 7, day 10, day 14,day 28).

SUMMARY:
This is a single cente, single arm, open-label, phase I study to evaluate the safety and effectiveness of CMV-TCR-T cell immunotherapy in treating CMV virus infection after HSCT.

DETAILED DESCRIPTION:
CMV infection is a common virus infection of HSCT, and which is highly related with the failure of transplantation and survival time of transplant patients. To evaluate the safety and efficacy of allogenic CMV-TCR-T cell therapy in subjects with CMV infection, patients with CMV emias or deseases will be enrolled, and donor derived CMV-TCR-T(HLA-A*1101\0201\2402) cells will be intravenously infused with a escalated dose of 0.1-1×106 CMV-TCR-T cells. The CMV DNA copies and CMV-TCR-T cell proliferation will be monitored in the scheduled time (day 0, day 4, day 7, day 10, day 14, day 28).

ELIGIBILITY:
Inclusion Criteria:

1. Age 1-70 years, including boundary values, gender unlimited;
2. Allogenic hematopoietic stem cell transplantation patients with CMV infection disease or persistent CMV emia;
3. At least one of the following conditions after allogeneic HSCT:

   * After trested with 2-week standard antiviral drug, compared to the baseline of treatment, the decrease of CMV DNA copies number was less than 1log10, and the CMV DNA copies number is greater than 1000 copies/ mL ;
   * Unable to tolerate the toxic and side effects of antiviral drugs,such as bone marrow hematopoietic suppression, nephrotoxicity;
4. Estimated life expectancy ≥3 months；
5. ECOG 3;
6. Patients who voluntarily sign informed consent and are willing to comply with treatment plans, visit arrangements, laboratory tests and other research procedures.

Exclusion Criteria:

1. Patients with active aGVHD III-IV and / or mild and severe cGVHD;
2. Received cell therapy such as DLI,CTL,CAR-T or participated in any other clinical study of drugs and medical devices before 30 days of enrollment.
3. Pregnant or lactating women;
4. Intracranial hypertension or confusion; respiratory failure; disseminated intravascular coagulation;
5. patients with organ failure:

   * Heart: NYHA heart function grade IV;
   * Liver: Grade C that achieves Child-Turcotte liver function grading;
   * Kidney: kidney failure and uremia;
   * Lung: symptoms of respiratory failure;
   * Brain: a person with a disability;
6. The researchers found that it was unsuitable for the recipients to be enrolled.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-12-19 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Percentage of adverse events | 3months
  Percentage of participants with adverse events.

SECONDARY OUTCOMES:
Persistence of TCR-T cells | 3months
Changes of CMV-DNA copies number | 3months

CONTACTS AND LOCATIONS:
Overall Officials: Xingyu Cao, Ph.D, Study Director — Hebei Yanda Ludaopei Hospital
Locations (1):
- Hebei Yanda Ludaopei Hospital, Sanhe, Hebei, China

REFERENCES:
- [Derived] Liu G, Chen H, Cao X, Jia L, Rui W, Zheng H, Huang D, Liu F, Liu Y, Zhao X, Lu P, Lin X. Efficacy of pp65-specific TCR-T cell therapy in treating cytomegalovirus infection after hematopoietic stem cell transplantation. Am J Hematol. 2022 Nov;97(11):1453-1463. doi: 10.1002/ajh.26708. Epub 2022 Sep 22. PMID 36054234